CLINICAL TRIAL: NCT02207010
Title: A Phase 0 Study of AZD1775 in Preoperative Glioblastoma Multiforme (GBM) Patients Scheduled for Resection to Evaluate for Central Nervous System (CNS) Penetration
Brief Title: A Phase 0 Study of AZD1775 in Recurrent GBM Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: The Ben & Catherine Ivy Foundation (Other); American Society of Clinical Oncology (Other); Barbara Ann Karmanos Cancer Institute (Other); Translational Genomics Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BBTRC 001
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Glioblastoma; GBM
Keywords: Glioblastoma; GBM; first recurrence
MeSH Terms: conditions — Glioblastoma | interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD1775 (Experimental): Patients will receive a single dose (either 100 mg, 200 mg or 400 mg) of AZD1775, an oral agent, prior to surgery for resection of GBM
  Interventions: Biological: AZD1775

INTERVENTIONS:
Biological: AZD1775 — All patients receive a single dose of the oral study drug prior to surgery for resection of GBM.
  Other Names: Wee1 inhibitor; MK1775

SUMMARY:
This study would test how much of the new drug, AZD1775, is present in tumor, blood, and skin after one dose of the drug.

The purpose of the study is not to treat the tumor, but to see if the drug actually gets into the tumor cells. This study does not replace routine cancer treatment.

DETAILED DESCRIPTION:
Patients will be administered one dose of AZD1775 prior to surgical resection of their tumor. There will be 2 portions of this trial, referred to as Part 1 and Part 2. Part 1 will involve a dose escalation strategy where 3 separate doses (100, 200, and 400mg) will be evaluated. Each dose cohort will involve 4 patients. Surgery, with tissue harvest for determination of both tissue drug level and biomarker evaluation, will occur at 8 hrs post drug administration.

Part 2 will determine the potential tumor drug level and PD effects at various time intervals after drug administration of a single select drug dose. Currently, we are planning to use a dose (200 mg) that has been deemed safe when used in combination with cytotoxic therapy. However, if results from Part 1 suggest an alternate dose may be preferable, we will consider using that alternate dose in Part 2. Dosing will be followed by surgical resection at 2-4 hrs and at 22-26 hrs post dose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with 1 prior resection of histologically-diagnosed de novo GBM
2. Patient must have MRI evidence of disease recurrence
3. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status ≤2
4. Patients ≥ 18 years of age
5. Adequate hematologic, renal, and hepatic function
6. Patients must not have co-morbid condition(s) that, at the opinion of the investigator, prevent safe surgical treatment
7. Patients must not have active infection or fever > 38.5°C
8. Patients must not be pregnant or nursing
9. Patients must have archival tumor tissue block available for research use
10. Ability to understand and the willingness to sign a written informed consent document.
11. Patient has voluntarily agreed to participate by giving written informed consent.

Exclusion Criteria:

1. Less than 18 years of age
2. Diagnosis of anything other than first-recurrence GBM
3. GBM tissue from first-resection not available
4. Previous treatment with AZD1775
5. Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
6. Patient has known hypersensitivity to the components of potential study therapy or its analogs.
7. Patient has had prescription or non-prescription drugs or other products known to be metabolized by cytochrome P450 3A4 (CYP3A4), or to inhibit or induce CYP3A4, which cannot be discontinued prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study medication (inhibitors generally for 5 half-lives). Medications of particular concern are the following inhibitors of CYP3A4: azole antifungals (ketoconazole itraconazole, fluconazole and voriconazole), macrolide antibiotics (erythromycin, clarithromycin), cimetidine, HIV protease inhibitors, nefazodone and the following inducers of CYP3A4: phenytoin, barbiturates and rifampicin. Substrates of CYP3A4 include statins (lovastatin, simvastatin), midazolam, terfenadine, astemizole, and cisapride. CYP3A4.
8. Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate.
9. Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
10. Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse.
11. Patients expecting to reproduce within the projected duration of the study (estimated to be 1 year), and women who are pregnant or breastfeeding.
12. Patient is known to be suffering from Acquired Immune Deficiency Syndrome (AIDS).
13. Patient has known history of Hepatitis B or C.
14. Patient has symptomatic ascites or pleural effusion. A patient who is clinically stable following treatment for these conditions is eligible.
15. Patient has a clinical history suggestive of Li-Fraumeni Syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of AZD1775 following single dose of AZD1775 | at baseline, 2-4, 8-12, and 22-26 hours following single dose of AZD1775
  Will be summarized using descriptive statistics
Intratumoral concentration of AZD1775 | up to day of surgery
  Will be summarized using descriptive statistics

SECONDARY OUTCOMES:
Degree of CDC2 (Tyr15) phosphorylation in tissue | at baseline and up to 26 hours post dosing
  Will be summarized using descriptive statistics
Number of GBM cells in M-phase of cell cycle (PH3) | at baseline and up to 26 hours post dose AZD1775
  Will be summarized using descriptive statistics
Presence of double-strand DNA damage (γH2AX). | at baseline and up to 26 hours post dose AZD1775
  Will be summarized using descriptive statistics

OTHER OUTCOMES:
P53 mutation status | up to time of surgery
  Will be summarized using descriptive statistics
Presence of checkpoint regulator genes in GBM specimens | up to time of surgery
  checkpoint regulator genes in GBM specimens

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Barrow Neurological Institute at St.Joseph's Hospital Medical Center
Locations (1):
- Barrow Neurological Institute at St. Joseph's Hospital Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Sanai N, Li J, Boerner J, Stark K, Wu J, Kim S, Derogatis A, Mehta S, Dhruv HD, Heilbrun LK, Berens ME, LoRusso PM. Phase 0 Trial of AZD1775 in First-Recurrence Glioblastoma Patients. Clin Cancer Res. 2018 Aug 15;24(16):3820-3828. doi: 10.1158/1078-0432.CCR-17-3348. Epub 2018 May 24. PMID 29798906